CLINICAL TRIAL: NCT01008514
Title: A Single Institution, Prospective, Non-randomized Study of Partial Breast Irradiation Using the MammoSite Radiation Therapy System (Breast Brachytherapy Applicator)
Brief Title: Partial-Breast Radiation Therapy in Treating Women With Early-Stage Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding issues and Principal Investigator leaving the institution
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08177
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: accelerated partial breast irradiation
Radiation: intracavitary balloon brachytherapy

SUMMARY:
RATIONALE: Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. It may also cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well partial-breast radiation therapy works in treating women with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To examine the efficacy of MammoSite® Radiation Therapy System (RTS) in delivering partial-breast irradiation to women with early-stage breast cancer.

Secondary

* To assess the toxicities associated with MammoSite® RTS in these patients.
* To evaluate the cosmetic results in the breast after brachytherapy with the MammoSite® RTS.
* To correlate the cosmetic results with the use of chemotherapy, volume of the implant, and distance from the implant to the skin.
* To correlate the local recurrence rate with time between surgery and implant.

OUTLINE: Patients undergo placement of the MammoSite® Radiation Therapy System (RTS) device into the cavity where the tumor was removed either at the time of surgery or percutaneously under ultrasound guidance after surgery. Within 2-5 days after the device implant, patients undergo partial-breast irradiation delivered by MammoSite® RTS twice daily for 5 days.

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS) of the breast or invasive breast adenocarcinoma

  * Stage 0, I, or II (T2, N0; tumor size ≤ 3 cm) disease
  * Pathologic staging of the axilla preferred

    * Clinical staging of the axilla allowed for patients ≥ 70 years of age with hormone receptor-positive tumors
* Unicentric tumor

  * Microscopic multifocality allowed as long as the total tumor size is ≤ 3 cm
* Must have undergone lumpectomy as definitive surgery

  * Negative surgical margins, defined as no tumor at the inked margin of resection after final surgery

    * Re-excision to obtain negative margins allowed
* Must have adequate skin spacing between balloon surface and surface of the skin and lung (≥ 7 mm)
* No multicentric carcinoma (invasive or DCIS) in more than one quadrant
* No clinically or pathologically positive regional lymph nodes
* No extensive intraductal component, defined as DCIS extending beyond the primary invasive component into normal breast parenchyma and composing > 25% of the primary tumor
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No collagen-vascular disease, including any of the following:

  * Dermatomyositis
  * Systemic lupus erythematosus
  * Scleroderma-mixed connective tissue disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Proportion of local recurrence | up to 5 years
  * Local recurrence is defined as either invasive or non-invasive local recurrence within the target volume.
  * Ipsilateral elsewhere recurrence is defined as either invasive or non-invasive local recurrence outside of the target volume.

SECONDARY OUTCOMES:
Safety and toxicity | up to 30 months after radiotherapy
Cosmetic results | up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu